CLINICAL TRIAL: NCT00164021
Title: The Prevalence and Significance of Gastro-oesophageal Reflux in Adults With Cystic Fibrosis Before and After Lung Transplantation, Together With the Effects of Physiotherapy Airway Clearance Techniques on Gastro-oesophageal Function
Brief Title: The Prevalence and Significance of Gastro-oesophageal Reflux in Cystic Fibrosis Before and After Lung Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bayside Health (Other Government)
Collaborators: The Alfred (Other); Monash University (Other)
Responsible Party: Sponsor
Other Study IDs: 1/01; Alfred Hospital $20,000 grant
Record Dates: First submitted 2005-09-13; First posted 2005-09-14 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Cystic Fibrosis
Keywords: gastroesophageal reflux, gastric reflux, acid reflux, lung transplantation, physiotherapy, anti-reflux medication
MeSH Terms: conditions — Cystic Fibrosis; Gastroesophageal Reflux | interventions — Physical Therapy Modalities; Exercise

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cystic Fibrosis: Patients with cystic fibrosis
  Interventions: Procedure: Physiotherapy, exercise, percutaneous gastrostomy feeds; Drug: Anti-reflux pharmacotherapy
- Control

INTERVENTIONS:
Procedure: Physiotherapy, exercise, percutaneous gastrostomy feeds
  Groups: Cystic Fibrosis
Drug: Anti-reflux pharmacotherapy
  Groups: Cystic Fibrosis

SUMMARY:
Gastro-oesophageal reflux (GOR) has been found to be prevalent in children with cystic fibrosis (CF)and may further worsen lung damage via reflex bronchospasm or pulmonary aspiration. Chest physiotherapy may result in increased episodes of GOR as demonstrated in children. Lung transplantation may worsen pre-existing GOR. This study will determine the prevalence, severity and significance of symptomatic and silent GOR in adults with CF before and after lung transplant using 24hr oesophageal pH monitoring, a valid symptom questionnaire, quality of life questionnaires and gastric emptying studies. This study will identify the extent of GOR in a large adult CF population and the impact on lung function and quality of life together with the effects of medical and physiotherapy treatment on gastro-oesophageal function.

DETAILED DESCRIPTION:
A factorial longitudinal study will be undertaken in adults with cystic fibrosis. Results will be compared with age matched healthy controls. It is not deemed appropriate to randomise patients with gastro-oesophageal reflux(GOR) to a treatment versus no treatment group as immediate treatment for GOR once diagnosed is regarded as obligatory.

Subjects: 180 adults with CF will be recruited from the Adult Cystic Fibrosis Unit at the Alfred Hospital to participate in the study. The ambulatory studies will be undertaken during baseline state in the outpatient setting. Fifteen age matched control subjects will be recruited from the general population.

Subjects who give their consent for participation in the study will undertake the following outcome measures:

1. Demographic data including age, gender, BMI, prescribed medication at the time of the study, lung function tests including FEV1, FVC, FEV1/FVC ratio and MMEF, genotype, pH of saliva and sputum.
2. Structured symptom questionnaire using a reliable valid measure developed by Carlsson et al 1998 will be used to assess patient's symptom scores.
3. Dual-channel 24hour oesophageal pH monitoring will be undertaken using a digitrapper (Medtronic, Sweden)and dual antimony tipped probe (Synectics, Sweden). Following calibration of the probes the distal antimony tip is positioned 5cm above the upper border of the lower oesophageal sphincter and the proximal probe 15 cm above the distal probe in the upper oesophagus.The patient will be instructed in using the three event buttons on the digitrapper recording start and finish time of meals, upright versus supine positioning and reflux episodes. The subject will be provided with a detailed 24hr 'Activity Diary' to record all meals (including percutaneous gastrostomy feeds), positions and activities including usual chest physiotherapy and physical exercise.The recorded pH information is downloaded into a computer program for analysis. The following indices will be measured in the distal and proximal oesophagus:

   * Number of reflux episodes
   * Fraction of reflux time
   * Number of reflux episodes with duration longer than 5 minutes
   * Duration of longest episodes in minutes
   * DeMeester score (an overall weighted score of gastro-oesophageal function).
4. Quality of life questionnaires: SF36, Quittner CF Questionnaire (CFQ), Dietary and Bowel Symptom Questionnaires.
5. Chest radiographs

ELIGIBILITY:
Inclusion Criteria:

* * Diagnosis of cystic fibrosis

  * Medically stable

Exclusion Criteria:

* * Known oesophageal varices

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients of the Cystic Fibrosis Unit
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2001-02; Primary Completion 2016-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Brenda M Button, DPhty, PhD, Principal Investigator — The Alfred; Susannah King, Principal Investigator — The Alfred; Colleen Ash, Principal Investigator — The Alfred; John W Wilson, MBBS, PhD, Principal Investigator — The Alfred; Greg Snell, MBBS, Principal Investigator — The Alfred; Stuart Roberts, MBBS, Principal Investigator — The Alfred
Locations (1):
- The Alfred Hospital, Melbourne, Victoria, Australia